CLINICAL TRIAL: NCT00935259
Title: A Randomized, Placebo Controlled Clinical Trial to Evaluate the Effects of Simvastatin Treatment on Measurements of Lipidomic Biomarkers in Men With Dyslipidemia
Brief Title: Lipid Biomarker Study in Men With Dyslipidemia After Simvastatin Treatment (Study MK-0000-140)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-140; 2009_609
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Results first posted 2012-02-20 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Hypercholesterolemia, Dyslipidemia
Keywords: Hypercholesterolemia, Dyslipidemia, simvastatin, Zocor
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin 40 mg first, then placebo (Experimental): Simvastatin 40 mg tablets once daily for 2 weeks followed by placebo for 2 weeks
  Interventions: Drug: Simvastatin; Drug: Placebo
- Placebo first, then simvastatin 40 mg once daily (Placebo Comparator): Placebo for 2 weeks followed by simvastatin 40 mg once daily for 2 weeks
  Interventions: Drug: Simvastatin; Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — 40 mg once daily for 2 weeks
  Other Names: Zocor
Drug: Placebo — Placebo, matching the simvastatin (40 mg) tablet as a single oral daily dose for 2 weeks

SUMMARY:
The purpose of this study was to provide human lipidomics standards with simvastatin treatment that were to be used for comparison with similar preclinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a Caucasian (including Hispanic) male
* Participant has a maximum waist size of 40 inches
* Participant does not currently use any lipid-altering medications
* Participant is in good health other than the diagnosis of dyslipidemia

Exclusion Criteria:

* Participant has had stomach ulcers within the last 3 months
* Participant has had a heart attack in the last 6 months or has angina
* Participant has chronic heart failure
* Participant has a history of stroke, seizures, or major neurological disorder
* Participant has a history of cancer
* Participant has a gastrointestinal condition that affects bowel movements
* Participant has type 1 or 2 diabetes

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

REFERENCES:
- [Derived] Chen F, Maridakis V, O'Neill EA, Hubbard BK, Strack A, Beals C, Herman GA, Wong P. The effects of simvastatin treatment on plasma lipid-related biomarkers in men with dyslipidaemia. Biomarkers. 2011 Jun;16(4):321-33. doi: 10.3109/1354750X.2011.561367. Epub 2011 Mar 21. PMID 21417623

RESULTS

PARTICIPANT FLOW:
Groups:
- Simvastatin 40 mg, Then Placebo: Simvastatin 40 mg once daily for 2 weeks followed by placebo once daily for 2 weeks
- Placebo First, Then Simvastatin 40 mg: Placebo once daily for 2 weeks followed by simvastatin 40 mg daily for 2 weeks
Period: Period 1
Arm/Group | Simvastatin 40 mg, Then Placebo | Placebo First, Then Simvastatin 40 mg
Started | 16 | 15
Completed | 15 | 14
Not Completed | 1 | 1
Not completed — Administrative (scheduling conflict) | 1 | 1
Period: Period 2
Arm/Group | Simvastatin 40 mg, Then Placebo | Placebo First, Then Simvastatin 40 mg
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All enrolled participants
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Arachidonic Acid Level After 2 Weeks of Treatment
Description: Arachidonic acid level (20:4n6) in the cholesterol ester lipid class.
  The mean reported was an adjusted mean, which was obtained from running a 2-period crossover model that had fixed treatment and period terms and a random participant term.
Time Frame: 2 weeks
Population: Only participants with complete arachidonic acid data were included.
Measure: Mean (Standard Deviation); unit: nmol
Groups:
- Simvastatin 40 mg: Simvastatin 40 mg once daily for 2 weeks followed by placebo once daily for 2 weeks
- Placebo: Placebo once daily for 2 weeks followed by simvastatin 40 mg daily for 2 weeks
Arm/Group | Simvastatin 40 mg | Placebo
Number analyzed (Participants) | 27 | 29
nmol | 259.1 (89.1) | 269.6 (85.2)
Statistical Analysis 1: Comparison: Simvastatin 40 mg vs Placebo; Test type: Superiority or Other; p = 0.455, Mixed Models Analysis — Endpoint was analyzed as appropriate for a 2-period crossover model using a mixed model with fixed terms of period and treatment with participants as a random factor; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = -10.4, Standard Deviation 52.1

2. Secondary Outcome: Fasting Blood Lipidomic Levels After 2 Weeks of Treatment
Description: Change in fasting blood cholesterol ester, lysophosphatidylcholine, phosphatidylcholine, phosphatidylethanolamine, and triacylglycerol levels compared to placebo.
  The mean reported was an adjusted mean.
Time Frame: 2 weeks
Population: Only participants with complete blood lipidomic data were included.
  For cholesterol ester 22:5n6, n=26 for the simvastatin arm and n=27 for the placebo arm.
Measure: Mean (Standard Deviation); unit: nmol
Groups:
- Simvastatin 40 mg: Simvastatin 40 mg once daily for 2 weeks followed by placebo for 2 weeks
- Placebo: Placebo once daily for 2 weeks followed by Simvastatin 40 mg once daily for 2 weeks
Arm/Group | Simvastatin 40 mg | Placebo
Number analyzed (Participants) | 27 | 29
nmol
  Cholesterol ester lipid 16:00 | 288.9 (102.1) | 345.1 (87.3)
  Cholesterol ester lipid 18:3n3 | 10.0 (4.8) | 14.4 (6.7)
  Cholesterol ester lipid 20:3n6 | 20.9 (10.5) | 23.5 (10.2)
  Cholesterol ester lipid 20:3n9 | 1.3 (1.1) | 1.2 (0.9)
  Cholesterol ester lipid 22:5n6 | 1.0 (0.8) | 1.1 (0.4)
  Cholesterol ester lipid 22:6n3 | 12.7 (5.1) | 14.8 (6.8)
  Lysophosphatidyl-choline lipid 20:4n6 | 11.1 (3.8) | 10.3 (2.7)
  Phosphatidyl-choline lipid 18:2n6 | 684.8 (224.9) | 824.9 (196.2)
  Phosphatidyl-choline lipid 20:3n6 | 117.4 (54.3) | 127.1 (58.8)
  Phosphatidyl-choline lipid 20:4n6 | 458.0 (138.4) | 443.2 (98.1)
  Phosphatidyl-choline lipid 22:5n3 | 30.3 (10.2) | 34.3 (12.8)
  Phosphatidyl-choline lipid 22:5n6 | 11.4 (6.4) | 12.1 (4.1)
  Phosphatidyl-ethanolamine lipid 18:2n6 | 21.8 (9.3) | 32.1 (15.5)
  Triacylglycerol 16:00 | 788.3 (431.6) | 1005.1 (662.2)
  Triacylglycerol 20:3n9 | 4.5 (5.5) | 4.9 (2.8)
Statistical Analysis 1: Comparison: Simvastatin 40 mg vs Placebo; Cholesterol Ester 16:00; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = -51.7
Statistical Analysis 2: Comparison: Simvastatin 40 mg vs Placebo; Cholesterol Ester 18:3n3; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = -4.5
Statistical Analysis 3: Comparison: Simvastatin 40 mg vs Placebo; Cholesterol Ester 20:3n6; Test type: Superiority or Other; p = 0.217, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = -2.5
Statistical Analysis 4: Comparison: Simvastatin 40 mg vs Placebo; Cholesterol Ester 20:3n9; Test type: Superiority or Other; p = 0.666, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = 0.1
Statistical Analysis 5: Comparison: Simvastatin 40 mg vs Placebo; Cholesterol Ester 22:5n6; Test type: Superiority or Other; p = 0.776, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = 0.0
Statistical Analysis 6: Comparison: Simvastatin 40 mg vs Placebo; Cholesterol Ester 22:6n3; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = -2.5
Statistical Analysis 7: Comparison: Simvastatin 40 mg vs Placebo; Lysophosphatidylcholine 20:4n6; Test type: Superiority or Other; p = 0.152, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = 1.1
Statistical Analysis 8: Comparison: Simvastatin 40 mg vs Placebo; Phosphatidylcholine 18:2n6; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = -132.1
Statistical Analysis 9: Comparison: Simvastatin 40 mg vs Placebo; Phosphatidylcholine 20:3n6; Test type: Superiority or Other; p = 0.325, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = -11.8
Statistical Analysis 10: Comparison: Simvastatin 40 mg vs Placebo; Phosphatidylcholine 20:4n6; Test type: Superiority or Other; p = 0.419, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = 18.3
Statistical Analysis 11: Comparison: Simvastatin 40 mg vs Placebo; Phosphatidylcholine 22:5n3; Test type: Superiority or Other; p = 0.070, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = -4.7
Statistical Analysis 12: Comparison: Simvastatin 40 mg vs Placebo; Phosphatidylcholine 22:5n6; Test type: Superiority or Other; p = 0.769, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = -0.2
Statistical Analysis 13: Comparison: Simvastatin 40 mg vs Placebo; Phosphatidylethanolamine 18:2n6; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = -11.1
Statistical Analysis 14: Comparison: Simvastatin 40 mg vs Placebo; Triacylglycerol 16:00; Test type: Superiority or Other; p = 0.016, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = -240.8
Statistical Analysis 15: Comparison: Simvastatin 40 mg vs Placebo; Triacylglycerol 20:3n9; Test type: Superiority or Other; p = 0.833, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = 0.1

3. Secondary Outcome: Serum Proprotein Convertase Subtilisin-like/Kexin Type 9 (PCSK9) Level
Description: Two days of standardized, pre-packaged meals were provided prior to the 10-hour fast required before blood collection. To assess how consumption of a meal would affect levels of plasma PCSK9, following each of the fasting blood draws, participants were asked to consume a high fat meal (heavy whipping cream + vanilla ice cream in a 1:4 ratio [dose = 162 g/m^2]) within 20 minutes. For the duration of the test, participants were to remain seated or recumbent until blood samples were drawn 4 h after meal completion.
  The mean reported was an adjusted mean (defined in first outcome measure).
Time Frame: 2 weeks
Population: Only participants with complete PCSK9 data were included.
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Simvastatin 40 mg | Placebo
Number analyzed (Participants) | 27 | 29
nmol
  Fed | 6.06 (2.34) | 4.69 (1.66)
  Fasted | 6.47 (2.11) | 5.51 (1.91)
Statistical Analysis 1: Comparison: Simvastatin 40 mg vs Placebo; Fasted; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = 0.90
Statistical Analysis 2: Comparison: Simvastatin 40 mg vs Placebo; Fed; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; An unstructured covariance and Kenward Roger degrees of freedom were assumed; Mean Difference (Final Values) = 1.40

4. Secondary Outcome: Blood Linoleic Acid Levels
Description: Change in blood linoleic acid levels for Cholesterol Ester compared to placebo.
Time Frame: 2 weeks
Population: Only participants with complete blood linoleic acid data were included.
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Simvastatin 40 mg | Placebo
Number analyzed (Participants) | 27 | 29
nmol | 1184.7 (393.4) | 1504.7 (327.8)

5. Secondary Outcome: Change in Fasting Delta 5 Desaturase Enzyme Activity Compared to Placebo
Description: Change in fasting delta 5 desaturase enzyme activity compared to placebo. Delta 5 desaturase enzyme activity is defined as the ratios of C20:4n-6 to C20:3n-6 and C20:5n-3 to C20:4n-3.
Time Frame: 2 weeks
Population: Only participants with complete fasting delta 5 desaturase enzyme activity data were included.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Simvastatin 40 mg | Placebo
Number analyzed (Participants) | 28 | 30
ratio
  Cholesterol ester c20:4n6 / c20:3n6 | 12.2234 (3.413) | 11.5662 (3.684)
  Cholesterol Ester c20:5n3/c20:4n3 | 17.9161 (7.738) | 16.3024 (9.465)
Statistical Analysis 1: Comparison: Simvastatin 40 mg vs Placebo; Cholesterol ester c20:4n6 / c20:3n6; Test type: Superiority or Other; p = 0.247, Mixed Models Analysis
Statistical Analysis 2: Comparison: Simvastatin 40 mg vs Placebo; Cholesterol ester c20:5n3 / c20:4n3; Test type: Superiority or Other; p = 0.151, Mixed Models Analysis

ADVERSE EVENTS:
Groups:
- Simvastatin: Simvastatin 40 mg tablets once daily for 2 weeks in either Period 1 or Period 2
- Placebo: Placebo to simvastatin tablets once daily for 2 weeks in either Period 1 or Period 2
Arm/Group | Simvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=30) | Placebo (N=30)
Tension headache (Nervous system disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications should include input from the investigator(s), and Sponsor personnel. Such input should be reflected in publication authorship. The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.